CLINICAL TRIAL: NCT01027702
Title: Phase I/II Study of Donor Lymphocyte Infusion With Methotrexate GVHD Prophylaxis to Hasten Immune Reconstitution After CD34+ Cell-Selected Transplant
Brief Title: Donor Lymphocyte Infusion After Alternative Donor Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor/ PI leaving institution, no plans to continue this research at this time
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCH BMT 09-02
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2017-10

CONDITIONS: Immunodeficiency
Keywords: Donor Lymphocyte Infusion; Immune Recovery; T cell depleted transplant; Mismatched related donor transplants; Unrelated donor transplants
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion of donor lymphocytes (Experimental): Patients will receive an infusion of donor lymphocyte after T-cell depleted transplant.
  Interventions: Biological: Infusion of donor lymphocytes

INTERVENTIONS:
Biological: Infusion of donor lymphocytes — A donor lymphocyte infusion will be given to provide T cells. There will be a dose escalation: 3 x 10^4, 4 x 10^4, 5 x 10^4, 6 X 10^4, 8 x 10^4, and 10 X10^4 cells/kg body weight. At least three patients will be assessed at each dose to determine safety before dose is increased.

SUMMARY:
The purpose of this study is to determine the ability of a donor lymphocyte infusion (DLI) given with methotrexate to hasten immune recovery without causing severe graft-versus-host disease (GVHD) in recipients who have had a T-cell depleted transplant.

DETAILED DESCRIPTION:
Studies have shown that giving donor T cells after a mismatched T cell-depleted stem cell transplant can speed up recovery of T cells in the patient. This approach can cause severe graft versus host disease (GVHD). The purpose of this study is to determine whether giving a donor lymphocyte infusion (DLI) with methotrexate can accelerate immune recovery in recipients of T cell-depleted stem cell transplants. Thirty days after a T-cell depleted transplant, patients will be given a DLI. They will be monitored for immune recovery as measured by CD4 count and for GVHD toxicity.

Patients will be separated into six cohorts based on dose of DLI received: 3 x 10^4, 4 x 10^4, 5 x 10^4, 6 X 10^4, 8 x 10^4, and 10 X10^4 cells/ kg of body weight. A minimum of 3 patients will be tested at each dose starting with the lowest dose. Dose escalation will continue until the dose associated with CD4 count >100 at Day +120 after transplant without significant GVHD is determined. All patients will receive thirteen doses of methotrexate after the DLI to prevent GVHD. Patients will be followed for 2 years for outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been treated on the LCH BMT 09-01 protocol
* Signed informed consent by patient or legal guardian

Exclusion Criteria:

* Active GVHD at the time when DLI are due
* History of acute GVHD > grade I prior to DLI
* Disease due to viral infection (eg. CMV) when DLI are due (asymptomatic viral replication or viral shedding is not a contraindication)
* Uncontrolled bacterial or fungal infection
* O2 saturation by pulse oximetry < 95%
* Bilirubin > 3mg/dL or ALT > 5 x upper limit of normal
* Creatinine > 3x baseline (at transplant)
* ANC (WBC x % neutrophils + bands) < 500/ul
* Significant effusions (eg. pleural or pericardial) or ascites
* EBV-related PTLD
* Persistent or increasing mixed chimerism requiring therapeutic DLI as defined on the LCH BMT 09-01 protocol

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gilman, MD, Principal Investigator — Department of Pediatrics, Levine Children's Hospital, Carolinas Healthcare System
Locations (1):
- Levine Children's Hospital, Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilman AL, Leung W, Cowan MJ, Cannon M, Epstein S, Barnhart C, Shah K, Hyland M, Fukes T, Ivanova A. Donor lymphocyte infusion and methotrexate for immune recovery after T-cell depleted haploidentical transplantation. Am J Hematol. 2018 Feb;93(2):169-178. doi: 10.1002/ajh.24949. Epub 2017 Nov 17. PMID 29047161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who received a CD34+ selected peripheral blood stem cell (PBSC) transplant on the companion study, LCH BMT 09-01, at Levine Children's Hospital between December 2009 and June 2016.
Pre-assignment Details: Subjects were enrolled to two cohorts based on donor type, Mismatched Related Donor (MMRD) and Matched Unrelated Donor (MUD).
Groups:
- MMRD: 3 x 10^4/kg DLI + MTX to Day +24: Mismatched Related Donor: Donor Lymphocyte Infusion (DLI) 3 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Day +1, +3, +10, +17, and +24
- MMRD: 3 x 10^4/kg DLI + MTX to Day +52: Mismatched Related Donor: Donor Lymphocyte Infusion (DLI) 3 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Days +1, +3, +10, +17, and +24, 7.5 mg/m2 on Days +31 and +38, 5 mg/m2 on days +45 and +52
- MMRD: 4 x 10^4/kg DLI + MTX to Day +52: Mismatched Related Donor: Donor Lymphocyte Infusion (DLI) 4 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Days +1, +3, +10, +17, and +24, 7.5 mg/m2 on Days +31 and +38, 5 mg/m2 on days +45 and +52
- MMRD: 4 x 10^4/kg DLI + MTX to Day +80: Mismatched Related Donor: Donor Lymphocyte Infusion (DLI) 4 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Days +1, +3, +10, +17, and +24, 7.5 mg/m2 on Days +31 and +38, 5 mg/m2 on days +45, +52, +59, +66, +73, and +80
- MMRD: 5 x 10^4/kg DLI + MTX to Day +80: Mismatched Related Donor: Donor Lymphocyte Infusion (DLI) 5 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Days +1, +3, +10, +17, and +24, 7.5 mg/m2 on Days +31 and +38, 5 mg/m2 on days +45, +52, +59, +66, +73, and +80
- MUD: 3 x 10^4/kg DLI + MTX to Day +24: Matched Unrelated Donor: Donor Lymphocyte Infusion (DLI) 3 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Day +1, +3, +10, +17, and +24
- MUD: 3 x 10^4/kg DLI + MTX to Day +52: Matched Unrelated Donor: Donor Lymphocyte Infusion (DLI) 3 x 10^4 cells/kg followed by methotrexate (MTX) 10 mg/m2 on Days +1, +3, +10, +17, and +24, 7.5 mg/m2 on Days +31 and +38, 5 mg/m2 on days +45 and +52
Period: Overall Study
Arm/Group | MMRD: 3 x 10^4/kg DLI + MTX to Day +24 | MMRD: 3 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +80 | MMRD: 5 x 10^4/kg DLI + MTX to Day +80 | MUD: 3 x 10^4/kg DLI + MTX to Day +24 | MUD: 3 x 10^4/kg DLI + MTX to Day +52
Started | 4 | 4 | 3 | 14 | 10 | 1 | 2
Completed | 3 | 2 | 2 | 10 | 9 | 1 | 1
Not Completed | 1 | 2 | 1 | 4 | 1 | 0 | 1
Not completed — Received subsequent therapy | 1 | 2 | 0 | 4 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infusion of Donor Lymphocytes
Number analyzed (Participants) | 38
Age, Customized [Number; unit: participants]
  < 1 year | 2
  1-2 years | 3
  2-4 years | 3
  4-6 years | 3
  6-8 years | 3
  8-10 years | 3
  10-12 years | 4
  12-14 years | 4
  14-16 years | 3
  16-18 years | 6
  > 18 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
  African American | 19
  Hispanic or Latino | 10
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immune Recovery Following Transplantation
Description: Immune recovery was measured by CD4+ cells > 100/μL by Day 120 following transplantation
Time Frame: 120 days after transplant
Population: Patients who received subsequent therapy, such as therapeutic DLI (eg. for treatment of viral infection or relapse), chemotherapy, or a PBSC infusion were considered not evaluable as this could interfere with response assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRD: 3 x 10^4/kg DLI + MTX to Day +24 | MMRD: 3 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +80 | MMRD: 5 x 10^4/kg DLI + MTX to Day +80 | MUD: 3 x 10^4/kg DLI + MTX to Day +24 | MUD: 3 x 10^4/kg DLI + MTX to Day +52
Number analyzed (Participants) | 3 | 2 | 2 | 10 | 9 | 1 | 1
Participants | 1 | 1 | 1 | 4 | 6 | 1 | 1
Statistical Analysis 1: Comparison: MMRD: 3 x 10^4/kg DLI + MTX to Day +24 vs MMRD: 3 x 10^4/kg DLI + MTX to Day +52 vs MMRD: 4 x 10^4/kg DLI + MTX to Day +52 vs MMRD: 4 x 10^4/kg DLI + MTX to Day +80 vs MMRD: 5 x 10^4/kg DLI + MTX to Day +80 vs MUD: 3 x 10^4/kg DLI + MTX to Day +24 vs MUD: 3 x 10^4/kg DLI + MTX to Day +52; This was a dose-escalation study to determine a target DLI dose at which the: 1. Probability of CD4+ cells > 100/µL by Day +120 is at least 66% and 2. Probability of grade II and III GVHD is at most 33%, probability of grade III GVHD is at most 17%, and no grade IV GVHD occurs Patients were assigned in cohorts of 3; Test type: Other; The study design consisted of two phases, a dose-escalation phase and a dose-confirmation phase. In the dose-escalation phase, patients were assigned in cohorts of 3. The dose escalation plan was: * If a grade IV acute GVHD event was observed at any dose, no more patients were assigned to this or higher dose levels unless the methotrexate dosing was modified. * If none of the initial three patients at a dose level experienced grade II/III GVHD and < 2/3 had a CD4+ count > 100 at Day +120, the next three patients were assigned to the next higher dose level. * If 1 out of 3 patients had grade III GVHD or 1 - 2 out of 3 patients had grade II GVHD and/or > 2/3 have a CD4+ count > 100 at Day +120, the dose was repeated for the next 3 patients. The dose of 5 x 10^4 CD3+ cells/kg was determined to be the optimal dose

2. Primary Outcome: Incidence and Severity of GVHD
Description: Patients were evaluated for acute GVHD due to prophylactic DLI between the day of prophylactic DLI infusion and Day +180 after transplant. GVHD was graded using standard criteria.
Time Frame: 180 days after transplant
Population: Patients that had not had grade II-IV acute GVHD following prophylactic DLI but received therapeutic DLI (eg. for treatment of viral infection or relapse), chemotherapy, or a PBSC infusion prior to Day +180 were considered not evaluable because these therapies may cause or prevent GVHD and affect the determination of this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | MMRD: 3 x 10^4/kg DLI + MTX to Day +24 | MMRD: 3 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +52 | MMRD: 4 x 10^4/kg DLI + MTX to Day +80 | MMRD: 5 x 10^4/kg DLI + MTX to Day +80 | MUD: 3 x 10^4/kg DLI + MTX to Day +24 | MUD: 3 x 10^4/kg DLI + MTX to Day +52
Number analyzed (Participants) | 3 | 2 | 2 | 10 | 9 | 1 | 1
Participants
  No GVHD/ Grade I GVHD | 2 | 1 | 1 | 9 | 8 | 1 | 1
  Grade II GVHD | 0 | 1 | 1 | 1 | 1 | 0 | 0
  Grade III/IV GVHD | 1 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: MMRD: 3 x 10^4/kg DLI + MTX to Day +24 vs MMRD: 3 x 10^4/kg DLI + MTX to Day +52 vs MMRD: 4 x 10^4/kg DLI + MTX to Day +52 vs MMRD: 4 x 10^4/kg DLI + MTX to Day +80 vs MMRD: 5 x 10^4/kg DLI + MTX to Day +80 vs MUD: 3 x 10^4/kg DLI + MTX to Day +24 vs MUD: 3 x 10^4/kg DLI + MTX to Day +52; [analysis description as in outcome 1, analysis 1]; Test type: Other; The study design consisted of two phases, a dose-escalation phase and a dose-confirmation phase. In the dose-escalation phase, patients were assigned in cohorts of 3. The dose escalation plan was: If a grade IV acute GVHD event was observed at any dose, no more patients were assigned to this or higher dose levels unless the methotrexate dosing was modified. If none of the initial three patients at a dose level experienced grade II/III GVHD and < 2/3 had a CD4+ count > 100 at Day +120, the next three patients were assigned to the next higher dose level. If 1 out of 3 patients had grade III GVHD or 1 - 2 out of 3 patients had grade II GVHD and/or > 2/3 have a CD4+ count > 100 at Day +120, the dose was repeated for the next 3 patients. The dose of 5 x 10^4 CD3+ cells/kg was determined to be the optimal dose

3. Secondary Outcome: Number of Participants With Infection and EBV-related Post-transplant Lymphoproliferative Disease (PTLD)
Description: Subjects were actively monitored for adenovirus, cytomegalovirus (CMV), human herpes virus 6 (HHV6), and Epstein-Barr virus (EBV) as part of standard post-transplant care. All infections were collected from date of DLI until 1 year after transplant.
Time Frame: 1 year
Population: Patients who relapsed and received subsequent chemotherapy were no longer followed for infections as these therapies increase the risk of infections.
Measure: Number; unit: participants
Arm/Group | Infusion of Donor Lymphocytes
Number analyzed (Participants) | 38
participants
  HHV-6 reactivation, no disease | 18
  Viral upper respiratory infections | 17
  Adenovirus reactivation, no disease | 11
  Clostridium difficile colitis | 9
  Sinusitis | 8
  CMV reactivation, no disease | 5
  Galactomannan positive | 5
  BK virus, no disease | 5
  BK virus, hemorrhagic cystitis | 4
  EBV-related lymphoproliferative disease | 4
  Bacteremia, gram negative | 4
  Herpes simplex virus | 4
  Bacteremia, gram positive | 4
  Acute otitis media | 3
  Candidiasis (non-invasive) | 3
  Pneumonia | 3
  Infection with normal ANC - grade 3 | 3
  Adenovirus disease | 2
  EBV reactivation, no disease | 2
  Varicella | 2
  Nocardia | 2
  Pneumonia- fungal | 1
  Methicillin-resistant staphylococcus aureus (MRSA) | 1
  Norovirus | 1
  Parvovirus B19 (low level) | 1
  Rotavirus | 1
  Sapovirus | 1
  Possible respiratory fungal infection (rhizomucor) | 1

ADVERSE EVENTS:
Time Frame: From the time of donor lymphocyte infusion (DLI) up to one year after transplant.
Description: Infections that met the definition of a Serious Adverse Event are reported as the type of infection, when the cause of infection was known.
Arm/Group | Infusion of Donor Lymphocytes
All-Cause Mortality (participants affected / at risk) | 12/38
Serious Adverse Events (participants affected / at risk) | 32/38
Other Adverse Events (participants affected / at risk) | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infusion of Donor Lymphocytes (N=38)
Fever (General disorders) | 24
HHV-6 reactivation (Infections and infestations) | 6
Graft vs Host disease (Immune system disorders) | 5
EBV-related lymphoproliferative disease (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/25
CMV reactivation (Infections and infestations) | 2
Infection w/ unknown absolute neutrophil count (ANC) (Infections and infestations) | 2
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 2
ALT/ AST elevated (Investigations) | 1
Infection- eye NOS (Infections and infestations) | 1
Pulmonary/ Upper Respiratory- other (Respiratory, thoracic and mediastinal disorders) | 1 — Blood tinged sputum following fungal pneumonia
BK virus/ hemorrhagic cystitis (Infections and infestations) | 1
Hypertension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Seizure (Nervous system disorders) | 1
Infection- select (Infections and infestations) | 1 — viral upper respiratory infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infusion of Donor Lymphocytes (N=38)
Neutropenia (Investigations) | 12 — grade 4
Platelet count decreased (Investigations) | 10
Leukopenia (Investigations) | 8 — grade 4
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/25
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 — grade 3
Rash (Skin and subcutaneous tissue disorders) | 4 — grade 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 — grade 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 — grade 4
ALT elevated (Metabolism and nutrition disorders) | 2 — grade 4
Hemorrage, GU- urinary NOS (Renal and urinary disorders) | 2 — Hemorrhagic cystitis
Hypertension (Vascular disorders) | 2 — grade 4
Hypokalemia (Metabolism and nutrition disorders) | 2 — grade 4
Pain (General disorders) | 2 — grade 3
Renal/ Genitorurinary NOS (Renal and urinary disorders) | 2 — grade 3
Seizures (Nervous system disorders) | 2 — grade 3
Lymphopenia (Investigations) | 3 — grade 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 — grade 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT01027702/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT01027702/ICF_001.pdf